CLINICAL TRIAL: NCT01664143
Title: A Single-Center, Randomized, Investigator/Subject-Blind, Multiple Ascending-Dose, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO5508887 Following Oral Administration in Healthy Subjects
Brief Title: A Single-Center Study of RO5508887 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: WP28102; 2012-000280-24 (EudraCT Number)
Record Dates: First submitted 2012-08-08; First posted 2012-08-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO5508887 (Experimental)
  Interventions: Drug: RO5508887

INTERVENTIONS:
Drug: Placebo — Multiple doses of placebo
  Arms: Placebo
Drug: RO5508887 — Multiple doses of RO5508887
  Arms: RO5508887

SUMMARY:
This single-center, randomized, double-blind, placebo-controlled study will evaluate the safety, pharmacokinetics and pharmacodynamics of RO5508887 in healthy volunteers. Volunteers will receive multiple-ascending doses of RO5508887 or matching placebo. The anticipated time on study treatment is 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, >/=18 years of age
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive
* Use of adequate contraception methods or surgically sterile

Exclusion Criteria:

* Evidence of active or chronic disease
* Regular consumption of drugs of abuse
* Regular smoker (>5 cigarettes per day)
* Infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV)
* History of significant allergic reactions
* Abnormal blood pressure
* Clinical significant abnormalities (e.g., cardiovascular, laboratory values)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of adverse events | 30 days

SECONDARY OUTCOMES:
Correlation of the age on pharmacokinetics of RO5508887 | 30 days
Correlation of the age on pharmacodynamics of RO5508887 | 30 days
Pharmacokinetics: plasma levels of RO5508887 | Predose and up to 144 hours post last dose, and at follow-up
Pharmacodynamics: Plasma levels of amyloid deposition markers | Predose and up to 144 hours post last dose
Correlation of the age on safety of RO5508887 | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France